CLINICAL TRIAL: NCT02785588
Title: Development of a MR Scanner Capable of Being Sited in a Neonatal Intensive Care Unit
Brief Title: Development of a MR Scanner Capable of Being Sited in a Neonatal Intensive Care Unit (Firefly Sheffield)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 114-2014-GES-0035
Record Dates: First submitted 2016-05-19; First posted 2016-05-30 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Neonatal Neuroimaging
Keywords: MRI Scanner; NICU

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3.0 T Neonatal MRI scanner (Other): All subjects who participate in this study will be scanned using the 3.0 T Neonatal MRI scanner.
  Interventions: Device: 3.0 T Neonatal MRI scanner

INTERVENTIONS:
Device: 3.0 T Neonatal MRI scanner — eligible subjects will undergo neonatal MRI scan procedure

SUMMARY:
This study investigates a novel magnetic resonance imaging (MRI) system designed by GEHC for imaging viable neonate and infant populations. This MR system has a smaller size and design features that may make it more feasible to locate the system in close proximity to care areas for neonates (birth - 1 month) and infants (>1 month to two years), such as clinical neonatal intensive care units (NICUs) and other infant and neonatal care departments.

DETAILED DESCRIPTION:
This study investigates a novel magnetic resonance imaging (MRI) system designed by GEHC for imaging viable neonate and infant populations. This MR system has a smaller size and design features that may make it more feasible to locate the system in close proximity to care areas for neonates (birth - 1 month) and infants (>1 month to two years), such as clinical neonatal intensive care units (NICUs) and other infant and neonatal care departments.

This is a two-phase prospective clinical study evaluating the performance and safety of the investigational MRI device for neonates and infants, including:

* Phase 1 - Initial feasibility assessment and optimization study (Phase 1) which may include hardware and software modifications. These studies are guided by a series of MR scanning procedures defined in sequential Sponsor-provided MR Procedure Documents
* Phase 2 - Controlled image and data collection study based on Phase 1 results, in which optimized scan procedure(s) according to MR Procedure Document(s) will be provided at the start of Phase 2 scanning and a fixed hardware and integrated software configuration will be applied for all subjects.

Investigator feedback on scanning conducted under each MR Procedure Document will be documented. Because the device is intended for use in viable neonate and infant populations, clinical data are required that cannot be conducted in any other populations or simulated on non-human models. Clinical images and associated data as well as assessments of image quality, workflow, and usability will be collected.

Images, associated image data, and subject data collected in both phases of this study may be used for future engineering development and activities that support MR product development, including Sponsor-authorized scientific and marketing activities. Summary evaluation of safety and performance from Phase 1 and Phase 2 may be used in support of regulatory submission, including filings for European CE mark.

ELIGIBILITY:
Inclusion Criteria:

* Currently admitted for treatment or observation at the investigational site at the time of enrolment;
* weight range less than 5.0 kg (<5.0 kg ) and more than 0.5 kg (>0.5 kg );
* Viable neonates (birth to 1 month of age) or infants (>1 month to two years of age);
* Able to safely undergo an MRI scan, as determined by medically qualified personnel;
* Have parent(s), guardian(s), or legally authorized representative(s) willing and able to provide written informed consent for the subject's participation;
* Are of appropriate size and shape to fit into the bore of the magnet, inclusive of all monitoring equipment, if any, necessary for the subject's routine clinical care based on standard of care measurement methods, in accordance with site policies :

  1. Maximum width (shoulder-to-shoulder measurement) less than eighteen (18 cm).
  2. Maximum length (head-to-foot measurement) less than sixty (60) cm.

Exclusion Criteria:

* Have parent(s), guardian(s), or legally authorized representative(s) that require that they accompany the subject into the MR environment that have contraindications to the MR environment or would otherwise be put at undue risk or discomfort, as determined by medically qualified personnel;
* Have any ferrous or electrical items or non-removable medical devices that are not compatible with MR scanning (including devices labelled as MR Unsafe, MR conditional for which the scanning conditions are not met, or without MR safety labelling that does not satisfy site MR safety requirements) that may pose hazards in the MR scanning or MR environment, in the opinion of the Principal Investigator or medically qualified personnel in accordance with the site's MR Safety policy;
* Have any contraindications or could otherwise be expected to experience detrimental effects to safety, well-being, or medical care, as determined by the Principal Investigator or medically qualified personnel in accordance with the site's MR Safety policy;
* Require any scheduled standard of care procedures that are expected to be adversely impacted by participation in this study, in the opinion of the principal investigator or medically qualified personnel; and
* Have been previously enrolled AND undergone any study procedures under the current study protocol (i.e. the same subject cannot undergo study procedures, including swaddling and/or MR scanning, more than once).

Ages: 1 Minute to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Griffiths, MD, PhD, Principal Investigator — University of Sheffield
Locations (1):
- University of Sheffield, Royal Hallamshire Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Phase 1: Initial Feasibility Assessment
Arm/Group | 3.0 T Neonatal MRI Scanner
Started | 49
Completed | 47
Not Completed | 2
Not completed — Breakdown of investigational device | 1
Not completed — Withdrawal by Subject | 1
Period: Phase2 Controlled Image &Data Collection
Arm/Group | 3.0 T Neonatal MRI Scanner
Started | 5 (Phase 2 participants represent newly enrolled participants.)
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There were 54 enrolled subjects, with 2 withdrawn, resulting in 52 completed subjects for Phases 1 and 2 together. Additionally, the data from these 2 withdrawn subjects were not included in any statistical analysis.
  Viable neonates and/or infant subjects that met inclusion criteria and did not meet exclusion criteria were included in this study.
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 52

OUTCOME MEASURES:

1. Primary Outcome: Image Diagnostic Quality for Phase 1
Description: Number of subject whose images were rated as Evaluable.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 47
Participants | 24

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event in Phase 1
Description: Safety will be assessed based on the number of Adverse Events in Phase 1.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 47
Participants | 1

3. Primary Outcome: Image Diagnostic Quality for Phase 2
Description: Number of subject whose images were rated as Evaluable.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 5
Participants | 5

4. Primary Outcome: Number of Participants Who Experienced an Adverse Event in Phase 2
Description: Safety will be assessed based on the number of Adverse Events in Phase 2.
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 5
Participants | 0

5. Secondary Outcome: Summary of Image Quality and Assessment for Phase 1
Description: Scores range from 1-Very Poor image quality to 5-Excellent image quality.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 47
score on a scale
  Overall Quality | 3.57 (0.773)
  Image Contrast | 3.85 (0.834)
  Presence Artifact | 3.02 (0.821)
  Signal to noise ratio | 3.72 (0.926)
  Tissue Contrast | 3.98 (0.766)
  Fat/Water Homogeneity | 3.64 (0.673)

6. Secondary Outcome: Summary of Image Quality and Assessments for Phase 2
Description: Scores range from 1-Very Poor image quality to 5-Excellent image quality.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 5
score on a scale
  Overall Quality | 4.2 (0.447)
  Image Contrast | 4.4 (0.548)
  Presence Artifact | 3.8 (0.447)
  Signal to noise ratio | 4 (0)
  Tissue Contrast | 4.2 (0.837)
  Fat/Water Homogeneity | 4 (0)

7. Secondary Outcome: Per Subject Workflow and Transport Information
Description: Summary of means and standard deviations.
Time Frame: 1 Day
Population: There were 54 enrolled subjects, with 2 withdrawn, resulting in 52 completed subjects for Phases 1 and 2 together. Additionally, the data from these 2 withdrawn subjects were not included in any statistical analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 52
minutes
  Time in sponsor swaddle | 66 (13.73)
  Entire procedure time | 66.33 (9.70)
  MRI Scan time | 35.15 (8.02)

8. Secondary Outcome: Overall Experience With the Neonatal MR Scanner Device Summary
Description: User survey results on a scale from 1 to 5, where 1 = strongly disagree and 5 = strongly agree.
  Question 1. I think that I would like to use this system frequently Question 2. I found the system unnecessarily complex Question 3. I thought the system was easy to use Question 4. I think that I would need support from a technician to be able to use this system Question 5. I found the various functions in this system were well integrated Question 6. I thought there was too much inconsistency in this system Question 7. I think that most people would learn to use this system very quickly Question 8. I found the system very cumbersome to use Question 9. I felt very confident using the system Question 10. I needed to learn a lot of things before I could get going with this system Question 11. I feel confident this system will meet my patient's needs Question 12. How likely is it that you would recommend this system to other professionals in your field?
Time Frame: 1 Day
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 52
score on a scale
  Question 1 | 4.13 (0.40)
  Question 2 | 1.77 (0.47)
  Question 3 | 4.25 (0.44)
  Question 4 | 1.90 (0.45)
  Question 5 | 4.02 (0.24)
  Question 6 | 2.17 (0.68)
  Question 7 | 4.20 (0.43)
  Question 8 | 1.73 (0.45)
  Question 9 | 4.12 (0.38)
  Question 10 | 1.88 (0.38)
  Question 11 | 4.06 (0.42)
  Question 12 | 4.15 (0.50)

9. Secondary Outcome: Bi-polar Product Description Scale
Description: A measure of bi-polar items (opposite items), rated on a scale from 1 to 7. Closer to 1 indicates a measure closer to the first item and closer to 7 indicates a measure closer to the second item.
Time Frame: 1 Day
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 52
score on a scale
  Learnable-Not Learnable | 1.25 (0.44)
  Inefficient-Efficient | 6.47 (0.50)
  Resistant-Responsive | 6.51 (0.61)
  Annoying-Pleasing | 6.22 (0.92)
  Satisfying-Dissatisfying | 1.92 (1.06)
  Ineffective-Effective | 6.25 (0.80)
  Fast-Slow | 1.57 (1.20)
  Unfamiliar-Familiar | 6.37 (0.63)
  Routine-Unusual | 1.65 (0.96)
  Easy-Difficult | 1.53 (0.70)
  Useful-Useless | 1.61 (0.78)
  Bad-Good | 6.51 (0.70)

10. Secondary Outcome: Technical Issues and Malfunctions
Description: Number and type of technical issues and device malfunctions
Time Frame: 1 Day
Population: as for outcome 7
Measure: Number; unit: number of occurrences
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 52
number of occurrences
  Technical Issues | 0
  Device Malfunction | 5

11. Secondary Outcome: Subject Change in Temperature
Time Frame: 1 Day
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | 3.0 T Neonatal MRI Scanner
Number analyzed (Participants) | 52
Degrees Celsius | 0.17 (0.23)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | 3.0 T Neonatal MRI Scanner
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 1/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.0 T Neonatal MRI Scanner (N=54)
Bradycardia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT02785588/Prot_SAP_000.pdf